CLINICAL TRIAL: NCT00071240
Title: The Use of Recombinant Growth Hormone to Enhance T-Cell Production in Adults Infected With HIV-1
Brief Title: Growth Hormone to Increase Immune Function in People With HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: The J. David Gladstone Institutes (Other); University of California, San Francisco (Other); National Center for Research Resources (NCRR) (NIH); EMD Serono (Industry)
Responsible Party: Laura A. Napolitano, M.D., Assistant Professor of Medicine, UCSF, Gladstone Institute of Virology and Immunology, UCSF
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R01AI043864 (NIH); R01AI043864 (NIH)
Record Dates: First submitted 2003-10-16; First posted 2003-10-17 (Estimated); Last update posted 2009-08-17 (Estimated); Status verified 2009-08

CONDITIONS: HIV Infections
Keywords: Growth Hormone; HIV; AIDS; Thymus; CD4 Cell; Immune System; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Human Growth Hormone; Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Growth Hormone Arm (Experimental): Growth hormone receipt in the first year, post-growth hormone follow-up in the second year
  Interventions: Drug: Somatropin (recombinant human growth hormone)
- 2 (Active Comparator): Observation only in the 1st year, GH receipt in the second year
  Interventions: Drug: Somatropin (recombinant human growth hormone)

INTERVENTIONS:
Drug: Somatropin (recombinant human growth hormone) — 3.0mg sc daily for 6 months, followed by 1.5mg sc daily for 6 months. Dose stopped, held or reduced by study investigators as indicated by adverse events
  Other Names: Serostim

SUMMARY:
Growth hormone plays an important role in the development of the immune system. Studies suggest that growth hormone may promote growth of the thymus, a gland responsible for the production of important immune cells called T cells. Since these cells are lost during the course of HIV infection, it is possible that growth hormone treatment could help restore the immune system. This study will determine whether the administration of growth hormone can increase the size and function of the thymus and cause an increase in the number of new T cells in the blood of people infected with HIV.

Study hypothesis: Growth hormone treatment will enhance T cell production in HIV infected adults.

DETAILED DESCRIPTION:
The thymus is the major organ of T cell production and is generally believed to be nonfunctional in adults. Even if nonfunctional, it is destroyed by HIV infection while T cells are destroyed in the peripheral lymphoid system. Given the absence of new T cell production and a pathologic acceleration of T cell destruction, the immune system collapses and immunodeficiency ensues.

However, some studies have demonstrated thymic function in adults with HIV disease. Such function may be induced by positive feedback regulation of T cell production and the presence or absence of such function may play a determinant role in disease progression and response to highly active antiretroviral therapy (HAART). These studies suggest that the thymus is functional in many adults with HIV disease and that thymic function might be induced as a consequence of HIV-mediated peripheral T cell depletion. Growth hormone is a potent regulator of thymic function. This study will determine whether true thymic function can be induced in HIV infected adults, whether such induction is indeed prompted by growth hormone, and whether thymic function plays a role in sustaining the T cell compartment in the face of peripheral T cell depletion.

Twenty-four volunteers will be enrolled in this 2 year study. All participants will receive 12 months of treatment with human growth hormone. Participants will be randomly assigned to one of two study arms. Twelve participants (Arm 1) will receive growth hormone during the first year of the study (3 mg given daily by subcutaneous injection, with dose reduction to 1.5 mg after 6 months). Twelve participants (Arm 2) will be enrolled in an observational control arm (no placebo injections) that will cross over to growth hormone treatment after 1 year. Participants, whether in Arm 1 or Arm 2, will have as many as 24 scheduled study visits during the 2 years after enrollment. In general, study visits occur every every 1 to 3 months. Study visits will include physical exams, blood tests, CT scans, PET scans, and DEXA scans.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* CD4 count 400 cells/mm3 or less
* HIV viral load less than 1000 copies/ml for 1 year prior to study entry; in some cases, viral load up to 5000 copies/ml will be acceptable
* Taking at least 2 anti-HIV medications

Exclusion Criteria:

* Diabetes
* Cancer. Patients with some cases of Kaposi's sarcoma or skin cancer will not be excluded.
* Some (not all) forms of heart disease
* Carpal Tunnel Syndrome
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2002-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Effect of 1 year of growth hormone treatment on thymus mass, naive and total T cells | Thymus mass- months 0,6,12; Naive and total T cells - months 1,3,6,9,12
TREC content in circulating lymphocytes | Months 0,1,3,6,9,12

SECONDARY OUTCOMES:
Effect of 1 year of growth hormone treatment on B cells, NK cells, CD34+ cells, activated T cells, circulating IGF-1 levels, circulating cytokine levels, T cell function and repertoire | T cell repertoire Months 0,6,12, all others Months 0,1,3,6,9,12
metabolic activity of thymus | Months 0, 12
body composition | Months 0,3,6,12

CONTACTS AND LOCATIONS:
Overall Officials: Laura A. Napolitano, MD, Principal Investigator — University of California, San Francisco; Joseph M. McCune, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Gladstone Institute of Virology and Immunology, San Francisco, California, United States

REFERENCES:
- [Background] Napolitano LA, Lo JC, Gotway MB, Mulligan K, Barbour JD, Schmidt D, Grant RM, Halvorsen RA, Schambelan M, McCune JM. Increased thymic mass and circulating naive CD4 T cells in HIV-1-infected adults treated with growth hormone. AIDS. 2002 May 24;16(8):1103-11. doi: 10.1097/00002030-200205240-00003. PMID 12004268
- [Result] Napolitano LA, Schmidt D, Gotway MB, Ameli N, Filbert EL, Ng MM, Clor JL, Epling L, Sinclair E, Baum PD, Li K, Killian ML, Bacchetti P, McCune JM. Growth hormone enhances thymic function in HIV-1-infected adults. J Clin Invest. 2008 Mar;118(3):1085-98. doi: 10.1172/JCI32830. PMID 18292808
- [Result] Tesselaar K, Miedema F. Growth hormone resurrects adult human thymus during HIV-1 infection. J Clin Invest. 2008 Mar;118(3):844-7. doi: 10.1172/JCI35112. PMID 18292816